CLINICAL TRIAL: NCT00987389
Title: Plasma Exchange and Glucocorticoid Dosing in the Treatment of Anti-neutrophil Cytoplasm Antibody Associated Vasculitis: an International Randomized Controlled Trial
Brief Title: Plasma Exchange and Glucocorticoids for Treatment of Anti-Neutrophil Cytoplasm Antibody (ANCA) - Associated Vasculitis
Acronym: PEXIVAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); University of Birmingham (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PEXIVAS; R01FD00351604 (Other Grant/Funding Number: Food and Drug Administration (FDA)); 2009-013220-24 (EudraCT Number); NCT03919825 (obsolete NCT alias)
Record Dates: First submitted 2009-09-23; First posted 2009-09-30 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Granulomatosis With Polyangiitis (Wegener's) (GPA); Microscopic Polyangiitis (MPA)
Keywords: Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Wegener's; ANCA-Associated Vasculitis; GPA; MPA; Treatment; Plasma exchange; Glucocorticoids; ANCA-Positive
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Vasculitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Plasma Exchange; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Plasma Exchange with Standard Glucocorticoids (Experimental): Participants in this arm undergo plasma exchange and take a standard glucocorticoid dose.
  Interventions: Procedure: Plasma Exchange; Drug: Glucocorticoids [Standard Dose]
- No Plasma Exchange with Standard Glucocorticoids (Active Comparator): Participants in this arm do not undergo plasma exchange and take a standard glucocorticoid dose.
  Interventions: Other: No Plasma Exchange; Drug: Glucocorticoids [Standard Dose]
- Plasma Exchange with Reduced-Dose Glucocorticoids (Experimental): Participants in this arm undergo plasma exchange and take a reduced glucocorticoid dose.
  Interventions: Procedure: Plasma Exchange; Drug: Glucocorticoids [Reduced Dose]
- No Plasma Exchange with Reduced-Dose Glucocorticoids (Active Comparator): Participants in this arm do not undergo plasma exchange and take a reduced glucocorticoid dose.
  Interventions: Other: No Plasma Exchange; Drug: Glucocorticoids [Reduced Dose]

INTERVENTIONS:
Procedure: Plasma Exchange — Plasma exchange is a procedure whereby blood is taken from the body and separated by a machine into blood cells and plasma, which is the liquid part of blood. The plasma is discarded and the blood cells are returned to the body with a plasma substitute.
  Arms: Plasma Exchange with Reduced-Dose Glucocorticoids; Plasma Exchange with Standard Glucocorticoids
Other: No Plasma Exchange — No plasma exchange.
  Arms: No Plasma Exchange with Reduced-Dose Glucocorticoids; No Plasma Exchange with Standard Glucocorticoids
Drug: Glucocorticoids [Standard Dose] — During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then the dose will decrease following a standard regimen.
  Arms: No Plasma Exchange with Standard Glucocorticoids; Plasma Exchange with Standard Glucocorticoids
Drug: Glucocorticoids [Reduced Dose] — During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then the dose will decrease following a reduced regimen.
  Arms: No Plasma Exchange with Reduced-Dose Glucocorticoids; Plasma Exchange with Reduced-Dose Glucocorticoids

SUMMARY:
The purpose of this study is to determine whether plasma exchange as well as immunosuppressive therapy are effective in reducing death and end-stage renal disease (ESRD). The trial will also study whether a reduced cumulative dosing regimen of glucocorticoids is as effective as a standard disease regimen.

The FDA-OOPD is one of the funding sources for this study.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (Wegener's) (WG) and microscopic polyangiitis (MPA) are syndromes of primary systemic vasculitis associated with anti-neutrophil cytoplasm antibodies (ANCA). Together, these syndromes are grouped as ANCA-associated systemic vasculitis (AAV).

Plasma exchange, a method of rapidly removing potentially pathogenic ANCA and other mediators of inflammation and coagulation, has shown promise as an adjunctive therapy in AAV to improve early disease control and improve rates of renal recovery in severe disease. Glucocorticoids (steroids) are a standard of care in the treatment of AAV. High doses of glucocorticoids early in disease, although reduce disease activity due to their anti-inflammatory and immunosuppressive properties, also increase the risk of infection, particularly in the elderly and in the presence of uremia. There is no randomized trial data to guide glucocorticoids dosing.

Patients with severe new or relapsing AAV and pulmonary hemorrhage and/or renal disease will be eligible for this trial.

Subjects participating in this study will be randomized to receive one of the following groups;

1. Plasma exchange - 7 exchanges and, either standard or low-dose glucocorticoids or
2. No plasma exchange and, either standard or low-dose glucocorticoids

All studies will receive standard remission-induction therapy with either cyclophosphamide or rituximab.

ELIGIBILITY:
Inclusion Criteria:

• New or previous clinical diagnosis of granulomatosis with polyangiitis or microscopic polyangiitis consistent with the Chapel-Hill consensus definitions

AND

• Positive test for proteinase 3-ANCA or myeloperoxidase-ANCA

AND

* Severe vasculitis defined by at least one of the following:

  1. Renal involvement characterized by both of the following:

     * Renal biopsy demonstrating focal necrotizing glomerulonephritis or active urine sediment characterized by glomerular haematuria or red cell casts and proteinuria

     AND
     * eGFR <50 ml/min/1.73 m2
  2. Pulmonary hemorrhage due to active vasculitis defined by:

     * A compatible chest x-ray or CT scan (diffuse pulmonary infiltrates)

     AND
     * The absence of an alternative explanation for all pulmonary infiltrates (e.g. volume overload or pulmonary infection)

     AND
  3. At least one of the following:

     * Evidence of alveolar hemorrhage on bronchoscopic examination or increasingly bloody returns with bronchoalveolar lavage
     * Observed hemoptysis
     * Unexplained anemia (<10 g/dL) or documented drop in hemoglobin >1 g/dL)
     * Increased diffusing capacity of carbon dioxide
* Provision of informed consent by patient or a surrogate decision maker

Exclusion Criteria:

* A diagnosis of vasculitis other than granulomatosis with polyangiitis or microscopic polyangiitis
* Positive serum anti-glomerular basement membrane antibody test or renal biopsy demonstrating linear glomerular immunoglobulin deposition
* Receipt of dialysis for >21 days immediately prior to randomization or prior renal transplant
* Age <15 years
* Pregnancy at time of study entry
* Treatment with >1 IV dose of cyclophosphamide and/or >14 days of oral cyclophosphamide and/or >14 days of prednisone/prednisolone (>30 mg/day) and/or >1 dose of rituximab within the 28 days immediately prior to randomization
* A comorbidity that, in the opinion of the investigator, precludes the use of cyclophosphamide, glucocorticoids, or plasma exchange or absolutely mandates the use of plasma exchange
* Plasma exchange in 3 months prior to randomization

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust; Peter Merkel, MD, MPH, Principal Investigator — University of Pennsylvania; Michael Walsh, MD, Principal Investigator — McMaster University
Locations (98):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Australia (18):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - John Hunter Hospital,, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Nambour Hospital, Nambour, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre,, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - The Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital,, Fremantle, Western Australia
  - Gold Coast Hospital, Southport
- University Hospitals Leuven, Leuven, Belgium
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - St Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Hopital Saint-Luc, Montreal, Quebec
- General Faculty Hospital, Prague, Czechia
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Holstebro Hospital and University of Aarhus, Holstebro
- France (17):
  - Centre Hospitalier de Boulogne, Boulogne-sur-Mer
  - CHRU Brest Hopital La Cavale Blanche, Brest
  - CHU Brest, Brest
  - CHU Caen - Nephrology Department, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Colmar Hospital - Nephrology, Colmar
  - CHU D'Angers, D'Angers
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hopital Site Sainte Blandine, Metz
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Cochin, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - Centre Hospitalier de la Region d'Annecy, Pringy
  - CHU De Toulouse-Hotel Dieu Saint Jacques, Toulouse
  - CHU Hopital Bretonneau, Tours
  - Centre Hospitalier de Valenciennes, Valenciennes
- Hippokration Hospital, Thessaloniki, Greece
- Italy (2):
  - University of Brescia, Brescia
  - Azienda Ospedaliero Universitaria di Parma, Parma
- Japan (6):
  - University of Tsukuba, Tsukuba, Ibaraki
  - Kyoto University Hospital, Kyoto
  - University of Miyazaki Hospital, Miyazaki
  - Kitano Hospital, Osaka
  - Teikyo University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico
- New Zealand (3):
  - North Shore Hospital, Takapuna, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Norway (2):
  - University Hospital North Norway HF, Tromsø
  - St Olavs Hospital, Trondheim University Hospital, Trondheim
- Sweden (3):
  - Linkoping University Hospital, Linköping
  - Skane University Hospital, Malmo
  - Karolinska Institute, Stockholm
- United Kingdom (21):
  - Western Infirmary, Glasgow, Scotland
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - Brighton and Sussex University Hospitals, Brighton
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon & Exeter Hospital (Wonford), Exeter
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Royal Free Hospital, London
  - The Royal London Hospital, London
  - St. George's Hospital, London
  - Hammersmith Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences, Oxford
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Royal Berkshire Hospital, Reading, Reading

REFERENCES:
- [Background] Walsh M, Merkel PA, Peh CA, Szpirt W, Guillevin L, Pusey CD, De Zoysa J, Ives N, Clark WF, Quillen K, Winters JL, Wheatley K, Jayne D; PEXIVAS Investigators. Plasma exchange and glucocorticoid dosing in the treatment of anti-neutrophil cytoplasm antibody associated vasculitis (PEXIVAS): protocol for a randomized controlled trial. Trials. 2013 Mar 14;14:73. doi: 10.1186/1745-6215-14-73. PMID 23497590
- [Result] Walsh M, Merkel PA, Peh CA, Szpirt WM, Puechal X, Fujimoto S, Hawley CM, Khalidi N, Flossmann O, Wald R, Girard LP, Levin A, Gregorini G, Harper L, Clark WF, Pagnoux C, Specks U, Smyth L, Tesar V, Ito-Ihara T, de Zoysa JR, Szczeklik W, Flores-Suarez LF, Carette S, Guillevin L, Pusey CD, Casian AL, Brezina B, Mazzetti A, McAlear CA, Broadhurst E, Reidlinger D, Mehta S, Ives N, Jayne DRW; PEXIVAS Investigators. Plasma Exchange and Glucocorticoids in Severe ANCA-Associated Vasculitis. N Engl J Med. 2020 Feb 13;382(7):622-631. doi: 10.1056/NEJMoa1803537. PMID 32053298
- [Derived] Fussner LA, Flores-Suarez LF, Cartin-Ceba R, Specks U, Cox PG, Jayne DRW, Merkel PA, Walsh M; PEXIVAS Investigators. Alveolar Hemorrhage in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis: Results of an International Randomized Controlled Trial (PEXIVAS). Am J Respir Crit Care Med. 2024 May 1;209(9):1141-1151. doi: 10.1164/rccm.202308-1426OC. PMID 38346237
- [Derived] Jayne D, Walsh M, Merkel PA, Peh CA, Szpirt W, Puechal X, Fujimoto S, Hawley C, Khalidi N, Jones R, Flossmann O, Wald R, Girard L, Levin A, Gregorini G, Harper L, Clark W, Pagnoux C, Specks U, Smyth L, Ito-Ihara T, de Zoysa J, Brezina B, Mazzetti A, McAlear CA, Reidlinger D, Mehta S, Ives N, Brettell EA, Jarrett H, Wheatley K, Broadhurst E, Casian A, Pusey CD. Plasma exchange and glucocorticoids to delay death or end-stage renal disease in anti-neutrophil cytoplasm antibody-associated vasculitis: PEXIVAS non-inferiority factorial RCT. Health Technol Assess. 2022 Sep;26(38):1-60. doi: 10.3310/PNXB5040. PMID 36155131
- See also: Related Info — http://www.rarediseasesnetwork.org/vcrc
- See also: Related Info — http://www.vasculitis.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 704 subjects were enrolled into the study and randomized to either plasma exchange or no plasma exchange, and randomized to receive either standard dose GC or reduced dose GC.
Groups:
- Plasma Exchange With Standard Glucocorticoids: Plasma Exchange: Plasma exchange is a procedure whereby blood is taken from the body and separated by a machine into blood cells and plasma, which is the liquid part of blood. The plasma is discarded and the blood cells are returned to the body with a plasma substitute.
  Glucocorticoids: During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then will follow a standard regimen.
- Plasma Exchange With Reduced Glucocorticoids: Plasma Exchange: Plasma exchange is a procedure whereby blood is taken from the body and separated by a machine into blood cells and plasma, which is the liquid part of blood. The plasma is discarded and the blood cells are returned to the body with a plasma substitute.
  Glucocorticoids: During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then the dose will decrease to a reduced regimen.
- No Plasma Exchange With Standard Glucocorticoids: Participants in this arm do not undergo plasma exchange.
  Glucocorticoids: During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then follow a standard regimen.
- No Plasma Exchange With Reduced Glucocorticoid: Participants in this arm do not undergo plasma exchange.
  All subjects' received the same glucocorticoids dose for the first two weeks, then the dose was decreased following a reduced glucocorticoid dose regimen.
Period: Overall Study
Arm/Group | Plasma Exchange With Standard Glucocorticoids | Plasma Exchange With Reduced Glucocorticoids | No Plasma Exchange With Standard Glucocorticoids | No Plasma Exchange With Reduced Glucocorticoid
Started | 176 | 176 | 175 | 177
Completed | 167 | 168 | 167 | 174
Not Completed | 9 | 8 | 8 | 3
Not completed — Ineligible | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 1
Not completed — Withdrawn from Treatment | 0 | 1 | 0 | 0
Not completed — Multiple different reasons | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- No Plasma Exchange: Participants in this arm do not undergo plasma exchange.
- Total: Total of all reporting groups
Arm/Group | Plasma Exchange | No Plasma Exchange | Total
Number analyzed (Participants) | 352 | 352 | 704
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (14.4) | 63.5 (13.7) | 63.2 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 158 | 307
  Male | 203 | 194 | 397
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  South Asian | 7 | 15 | 22
  Arab | 0 | 1 | 1
  Chinese | 1 | 5 | 6
  Japanese | 6 | 6 | 12
  Other Asian | 0 | 2 | 2
  Black African | 4 | 2 | 6
  Coloured African | 0 | 1 | 1
  Other Black | 5 | 2 | 7
  European | 281 | 277 | 558
  Latin America | 5 | 5 | 10
  Native N/S American or Aborigine | 16 | 7 | 23
  Other | 24 | 28 | 52
  Missing | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 15 | 39
  Czechia | 7 | 3 | 10
  Japan | 6 | 6 | 12
  United Kingdom | 88 | 91 | 179
  New Zealand | 6 | 4 | 10
  Canada | 97 | 94 | 191
  Sweden | 5 | 4 | 9
  Belgium | 1 | 0 | 1
  Norway | 0 | 8 | 8
  Denmark | 25 | 32 | 57
  Italy | 18 | 8 | 26
  Mexico | 4 | 3 | 7
  Australia | 44 | 50 | 94
  France | 21 | 31 | 52
  Poland | 5 | 2 | 7
  Spain | 1 | 1 | 2
ANCA Binding Specificity: PR3 [Count of Participants; unit: Participants] | 143 | 143 | 286
ANCA Binding Specificity: MPO [Count of Participants; unit: Participants] | 209 | 209 | 418
Severity of Renal Disease at Presentation: Creatinine <500umol/min [Count of Participants; unit: Participants] | 251 | 248 | 499
Severity of Renal Disease at Presentation: Requiring Dialysis or Creatinine >=500umol/min [Count of Participants; unit: Participants] | 101 | 104 | 205

OUTCOME MEASURES:

1. Primary Outcome: Composite of i) All-cause Mortality or ii) End-stage Renal Disease
Description: The primary outcome was a composite of death from any cause or end-stage renal disease (ESRD), defined as ≥12 continuous weeks of renal replacement therapy.
Time Frame: Time frame varied by subject: minimum of 1 year - maximum of 7 years
Measure: Count of Participants; unit: Participants
Groups:
- Plasma Exchange: Plasma Exchange: Plasma exchange is a procedure whereby blood is taken from the body and separated by a machine into blood cells and plasma, which is the liquid part of blood. The plasma is discarded and the blood cells are returned to the body with a plasma substitute.
  Glucocorticoids: During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then the dose will decrease following either a standard regimen or a reduced regimen.
- No Plasma Exchange: Participants in this arm do not undergo plasma exchange
  Glucocorticoids: During the study, a standard glucocorticoids dose regimen will be compared to a reduced glucocorticoids dose regimen. All subjects' patients will receive the same glucocorticoids dose for the first two weeks then the dose will decrease following either a standard regimen or a reduced regimen.
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
Participants | 100 | 109

2. Secondary Outcome: Number of Participants With Sustained Remission
Description: Remission that occurs before 6 months, and lasts without a first relapse until at least 12 months after randomization
Time Frame: Time frame varied by subject: minimum of 1 year - maximum of 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
Participants | 200 | 197

3. Secondary Outcome: Rate of Serious Infection Events
Description: Serious infections defined as an infectious syndrome that requires intravenous antibiotics or hospitalization for treatment.
Time Frame: Time frame varied by subject: minimum of 1 year - maximum of 7 years
Measure: Number; unit: events
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
events | 145 | 132

4. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: Quality of life was measured using the 36-item Short Form (SF-36) physical composite scores. Scores for the scale range from 0-100 and transformed to have a mean of 50 and SD of 10 in the reference population, with higher scores indicating a better Health-related Quality of Life.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Plasma Exchange: Participants in this arm undergo plasma exchange and take take either a standard glucocorticoid dose or a reduced glucocorticoid dose.
  Plasma Exchange: Plasma exchange is a procedure whereby blood is taken from the body and separated by a machine into blood cells and plasma, which is the liquid part of blood. The plasma is discarded and the blood cells are returned to the body with a plasma substitute.
- No Plasma Exchange: Participants in this arm do not undergo plasma exchange and take either a standard glucocorticoid dose or a reduced glucocorticoid dose.
  No Plasma Exchange: No plasma exchange.
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
units on a scale | 39.04 [38.58 to 41.65] | 37.96 [37.5 to 40.57]

5. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: Quality of life was measured using the 36-item Short Form (SF-36) mental composite scores. Scores for the scale range from 0-100 and transformed to have a mean of 50 and SD of 10 in the reference population, with higher scores indicating a better Health-related Quality of Life.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
score on a scale | 51.94 [51.27 to 53.70] | 51.40 [50.73 to 53.16]

6. Secondary Outcome: Health-related Quality of Life Using the EQ-5D Index Descriptive System
Description: EuroQoL-5 Dimensions consist of 2 elements: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprised of following 5 dimensions: 1.Mobility, 2.Self-Care, 3.Usual Activities, 4.Pain/Discomfort and 5.Anxiety/Depression. Each of these 5 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The digits for each of 5 dimensions were combined in a 5-digit number describing the participant's health state: e.g. state 11111 indicates no problem on any of the 5 dimensions. Health state index scores generally range from less than 0 (where 0 is a health state equivalent to death; negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating higher health utility.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Plasma Exchange | No Plasma Exchange
Number analyzed (Participants) | 352 | 352
score on a scale | 0.79 [0.78 to 0.84] | 0.77 [0.76 to 0.82]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of consent through study completion. The first subject was enrolled in June 2010, and the study completed in July 2017. Adverse event data was collected for 7 years and 1 month.
Arm/Group | Plasma Exchange | No Plasma Exchange
All-Cause Mortality (participants affected / at risk) | 46/352 | 53/352
Serious Adverse Events (participants affected / at risk) | 225/352 | 224/352
Other Adverse Events (participants affected / at risk) | 0/352 | 0/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma Exchange (N=352) | No Plasma Exchange (N=352)
Cardiovascular (Cardiac disorders) | 69 | 55
Endocrine (Endocrine disorders) | 9 | 2
Gastrointestinal (Gastrointestinal disorders) | 34 | 39
Hematological (Blood and lymphatic system disorders) | 25 | 16
Infection (Infections and infestations) | 136 | 114
Renal (Renal and urinary disorders) | 41 | 36
Surgery (Vascular disorders) | 16 | 13
Vasculitis Relapse (Immune system disorders) | 23 | 32
Other (General disorders) | 89 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT00987389/Prot_SAP_000.pdf